CLINICAL TRIAL: NCT04507750
Title: A Single-arm, Prospective Clinical Study of Camrelizumab Combined With Apatinib Mesylate in the Treatment of Relapsed Platinum-resistant Epithelial Ovarian Cancer
Brief Title: Camrelizumab Combined With Apatinib in the Treatment of Epithelial Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jing Liang, Professor, Qianfoshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYLL-KY-2020-(028)
Record Dates: First submitted 2020-07-30; First posted 2020-08-11 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Immune Checkpoint Inhibition
Keywords: camrelizumab; apatinib
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- camrelizumab+apatinib mesylate (Experimental): Carmelizumab: Intravenous infusion of a fixed dose of 200 mg in 30 minutes (not less than 20 minutes, not more than 60 minutes), once every 3 weeks, continuous administration until the disease progresses, the patient If death or intolerable toxicity occurs, medication for up to 1 year; Apatinib mesylate tablets: The initial dose is 250 mg, administered once a day, and continue to be administered. If there is a grade 3 to 4 adverse reaction, it should be administered once every other day.
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Carmelizumab: Intravenous infusion of a fixed dose of 200 mg in 30 minutes (not less than 20 minutes, not more than 60 minutes), once every 3 weeks, continuous administration until the disease progresses, the patient If death or intolerable toxicity occurs, medication for up to 1 year; Apatinib mesylate tablets: The initial dose is 250 mg, administered once a day, and continue to be administered. If there is a grade 3 to 4 adverse reaction, it should be administered once every other day.
  Other Names: apatinib mesylate

SUMMARY:
The aim of this study is to explore the effectiveness and safety of camrelizumab combined with apatinib mesylate in the treatment of relapsed platinum-resistant epithelial ovarian cancer

DETAILED DESCRIPTION:
The anti-PD-1 drug camrelizumab combined with apatinib mesylate was used to treat relapsed platinum-resistant epithelial ovarian cancer, and the effectiveness and safety of the treatment plan was evaluated by objective remission rate, progression-free survival, and major safety indicators , so as to provide patients a more beneficial treatment plan.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18 to 80 years old;

  2. Histologically diagnosed as epithelial ovarian cancer, fallopian tube cancer, and primary peritoneal cancer;

  3. Have received at least two lines of systemic chemotherapy;

  4. Platinum resistance (disease progression occurs within 6 months after the last platinum-containing chemotherapy Development) or platinum refractory (disease progression during platinum-containing chemotherapy), ovarian cancer,Fallopian tube cancer, primary peritoneal cancer;

  5. There are measurable lesions (according to RECIST 1.1 standard tumor lesion CT scan long diameter≥10mm, CT scan of lymph node lesions (short diameter≥ 10mm);

  6. ECOG score: 0-1 points;

  7. Estimated survival period ≥ 3 months;

  8. The main organs function well, and the inspection indicators meet the following requirements:Routine blood examination: hemoglobin ≥90 g/L (no blood transfusion within 14 days); neutrophil count ≥1.5×109/L; platelet count ≥80×109/L; biochemical examination: total bilirubin ≤1.5×ULN ( Upper limit of normal); alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤ 2.5×ULN; if there is liver metastasis, ALT or AST ≤ 5×ULN; endogenous creatinine clearance ≥ 50 ml/min (Cockcroft -Gault formula);

  9. The main organs are functioning normally, no blood transfusion or blood products within 14 days;

  10. Subjects of childbearing age must agree to take effective contraceptive measures during the trial;Age women's serum or urine pregnancy test must be negative; non-lactating patients;

  11. Subjects voluntarily join the study and sign an informed consent form, with good compliance and matchingClose follow-up.

Exclusion Criteria:

* 1. The subject has any active autoimmune disease or a history of autoimmune disease;

  2. Severe allergic reaction to other monoclonal antibodies;

  3. Suffer from other malignant tumors at the same time, except for malignant tumors that have been cured or have stable disease;

  4. The subject has previously received anti-PD-1, anti-PD-L1, anti-CD137 or anti-cytotoxic T lymphocyte-associated antigen-4 (CTLA-4) antibodies (including ipilimumab or any other specific targeting T cell Co-stimulation or checkpoint pathway antibodies or drugs) treatment;

  5. Pregnant or breastfeeding women;

  6. Patients who have used anti-angiogenesis therapy in the past, including bevacizumab, apatinib, or anlotinib;

  7. Participated in other drug clinical trials within three months;

  8. There are many factors that affect oral medications (such as inability to swallow, chronic diarrhea, ulcerative colitis and intestinal obstruction, etc.);

  9. Any bleeding event with a severity level of CTCAE4.0 or higher in the 4 weeks before screening;

  10. Patients with known central nervous system metastasis or a history of central nervous system metastasis before screening;

  11. Patients with hypertension who cannot be well controlled by a single antihypertensive drug treatment (systolic blood pressure> 140 mmHg, diastolic blood pressure> 90 mmHg); people with a history of unstable angina; a new diagnosis of angina within 3 months before screening Patients or myocardial infarction events occurred within 6 months before screening; Arrhythmia (including QTcF) requires long-term use of antiarrhythmic drugs and New York Heart Association grade ≥ Grade II cardiac insufficiency;

  12. Long-term unhealed wounds or fractures with incomplete healing;

  13. Have a history of organ transplantation;

  14. Imaging shows that the tumor has invaded important blood vessels or the researcher has judged that the patient's tumor is highly likely to invade important blood vessels and cause fatal bleeding during treatment;

  15. Abnormal coagulation function (PT>16s, APTT>43s, TT>21s, Fbg<2g/L), those with bleeding tendency (14 days before randomization must meet: INR is normal without using anticoagulants Within the range of values); patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin or their analogs; on the premise of prothrombin time international normalized ratio (INR) ≤ 1.5, use for preventive purposes is permitted Low-dose warfarin (1 mg orally, once a day) or low-dose aspirin (do not exceed 100 mg per day);

  16. Arterial/venous thrombosis events occurred in the year before screening, such as cerebrovascular accidents (including temporary ischemic attacks), deep vein thrombosis (venous thrombosis caused by intravenous catheterization due to pre-chemotherapy, except those who have been cured by the investigator ) And pulmonary embolism;

  17. People with a history of psychotropic drug abuse and unable to quit or have mental disorders;

  18. According to the judgment of the investigator, there are concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study.

  19. Live vaccines may be vaccinated during the study period less than 4 weeks before the study medication;

  20. Other researchers believe that it is not suitable for inclusion.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-08-10 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | within 1 year
  the proportion of patients with tumor size reduction of a predefined amount

SECONDARY OUTCOMES:
Progression Free Survival | within 1 year
  the length of time during and after the treatment of a disease, such as cancer, that a patient lives with the disease but it does not get worse
Disease Control Rate | within 1 year
  Refers to the percentage of confirmed complete remission, partial remission and stable disease (≥ 8 weeks) among patients with evaluable efficacy.
drug safety | within 1 year
  Incidence of test drug relative adverse events,Incidence of serious adverse events
6 months and 12 months overall survival | within 2 year
  It is the percentage of people in a study or treatment group still alive for a given period of time after diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Liang Jing, doctor, Principal Investigator — Qianfoshan Hospital
Locations (1):
- Shandong Provincial Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No